CLINICAL TRIAL: NCT01742741
Title: Early Feasibility Study 2 of Outpatient Control-to-Range - Testing System Efficacy (France)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Padova (Other); University of California, Santa Barbara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: France; JDRF 22-2011-649 (Other Grant/Funding Number: Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1 (T1DM); Continuous Glucose Monitor (CGM); Artificial Pancreas (AP); Insulin Pump; Closed Loop Control (CLC); Open Loop treatment; Diabetes Assistant; DiAs
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Involving Automated CTR (Experimental): Closed-Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs)system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct the hyperglycemia. The total doses recommended by the DiAs prior to meals and snacks includes the correction dose and Insulin on Board (IOB) calculated by the system.
  Interventions: Device: Diabetes Assistant (DiAs)
- CGM-Augmented Insulin Pump Treatment (No Intervention): Open Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in open-loop mode. Subjects will interact with the system through its Graphic User Interface (GUI). Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings. Subjects will be reminded that all treatment decisions should be based on fingerstick values and not on continuous glucose monitor (CGM) values.

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) — A medical platform that uses a smart-phone to connect to a continuous glucose sensor to insulin pump and run closed-loop control. The cell phone runs the Control to Range and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range (80-180 mg/dL during the day) and help avoid hypoglycemia during the night.
  Arms: Experimental Involving Automated CTR

SUMMARY:
An unblinded, randomized, cross-over design with each patient participating in two 40-hour outpatient admissions: (a) Experimental involving automated Control-to-Range (CTR) and (b) Control using Continuous Glucose Monitor (CGM)-augmented insulin pump treatment outside of a hospital based clinical research center.

DETAILED DESCRIPTION:
The principal goal is to validate a smart phone-based control-to-range (CTR) system for ambulatory use and to estimate the effect of CTR vs. sensor-augmented pump therapy, thereby providing justification for further larger home-based trials of CTR.

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 and <65 years old.
2. Clinical diagnosis of type 1 diabetes mellitus. For an individual to be enrolled at least one criterion from each list must be met.

   o Criteria for documented hyperglycemia (at least 1 must be met): i. Fasting glucose ≥126 mg/dL - confirmed ii. Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL - confirmed iii. HbA1c ≥6.5% documented - confirmed iv. Random glucose ≥200 mg/dL with symptoms v. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

   o Criteria for requiring insulin at diagnosis (1 must be met): i. Participant required insulin at diagnosis and continually thereafter ii. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually iii. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year.
4. Familiarity with a bolus calculator with the current insulin pump with pre-defined parameters for carbohydrate (CHO) ratio, insulin sensitivity factor (ISF), target glucose and active insulin.
5. HbA1c <9% as measured with DCA2000 or equivalent device.
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females).
7. Demonstration of proper mental status and cognition for the study.
8. Willingness to avoid consumption of acetaminophen-containing products during the study interventions involving CGM use.
9. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study.

Exclusion Criteria:

1. Severe hypoglycemia resulting in seizure, loss of consciousness, or diabetic ketoacidosis within the 12 months prior to enrollment.
2. Pregnancy; breast feeding, or intention of becoming pregnant.
3. Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg).
4. Conditions which may increase the risks associated with possible hypoglycemia, such as any active cardiac disorder/arrhythmia, uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation.
5. Self-reported hypoglycemia unawareness.
6. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans.
7. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants).
8. Anticoagulant therapy other than aspirin.
9. Oral steroids.
10. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
11. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment).
12. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
13. Known current or recent alcohol or drug abuse.
14. Medical conditions that would make operating a CGM, the DiAs cell phone or insulin pump difficult (e.g. blindness, severe arthritis, immobility).
15. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis).
16. In adherence with the One Touch Ultra 2 User Guide, subjects with hematocrit levels less than 30% and above 55% will be excluded.
17. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥three times the upper reference limit.
18. Impaired renal function measured as creatinine >1.2 times above the upper limit of normal.
19. Uncontrolled microvascular (diabetic) complications, such as current proliferative diabetic retinopathy or macular edema, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment.
20. Active gastroparesis requiring current medical therapy.
21. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study.
22. Uncontrolled thyroid disease.
23. Known bleeding diathesis or dyscrasia.
24. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor.
25. Active enrollment in another clinical trial.
26. Use of anti-diabetic agents other than continuous subcutaneous insulin infusion (CSII) including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, DPP-IV inhibitors, glucagon-like peptide 1 agonists, and alpha-glucosidase inhibitors
27. Subjects with basal rates less than 0.01U/hr.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Effect size of Control-to-Range (CTR) vs. Continuous Glucose Monitor (CGM)-augmented insulin pump treatment in an outpatient setting. | 40 hours
  The investigators expect that compared to CGM-augmented insulin pump treatment, CTR will result in moderate effect size of approximately 0.4, in terms of reduction of the overnight risk for hypoglycemia as measured by the Low Blood Glucose Index computed from retrofitted CGM data. This effect is not expected to be statistically significant with the anticipated sample size but will be used to inform power analysis for the subsequent multi-center trial of CTR at home.

SECONDARY OUTCOMES:
Time spent in target range | 40 hours
  CTR will improve (non-significantly at the projected sample size of N=5 subjects/site) the time spent within the target range of 80-140 mg/dL overnight (computed from retrofitted CGM data) and will reduce the extent of postprandial glucose excursions during the day. These data will provide justification and design support for a subsequent larger multi-center trial of CTR at home.

OTHER OUTCOMES:
Patient comfort with the Diabetes Assistant (DiAs) user interface | 40 hours
Reliability of DiAs remote monitoring | 40 hours
  Assess the DiAs remote monitoring by medical personnel/technicians to confirm appropriate functioning outside of the hospital setting.
Reliability of inter-device connections between DiAs and the CGM and between DiAs and the insulin pump. | 40 hours
  Assess the functioning of the connections between DiAs, the continuous glucose sensor, and the insulin pump.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Renard, MD, PhD, Principal Investigator — University of Montpellier Hospital; Boris P. Kovatchev, PhD, Study Director — University of Virginia
Locations (1):
- Centre d'Investigation Clinique CHU Montipellier, Montpellier, France

REFERENCES:
- [Derived] Kovatchev BP, Renard E, Cobelli C, Zisser HC, Keith-Hynes P, Anderson SM, Brown SA, Chernavvsky DR, Breton MD, Mize LB, Farret A, Place J, Bruttomesso D, Del Favero S, Boscari F, Galasso S, Avogaro A, Magni L, Di Palma F, Toffanin C, Messori M, Dassau E, Doyle FJ 3rd. Safety of outpatient closed-loop control: first randomized crossover trials of a wearable artificial pancreas. Diabetes Care. 2014 Jul;37(7):1789-96. doi: 10.2337/dc13-2076. Epub 2014 Jun 14. PMID 24929429